CLINICAL TRIAL: NCT02345044
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Study to Evaluate Efficacy and Safety of CS-3150 in Japanese Subjects With Hypertension
Brief Title: A Study to Evaluate Efficacy and Safety of CS-3150 in Japanese Hypertensive Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS3150-A-J203
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Essential Hypertension
Keywords: Essential hypertension; mineralocorticoid receptor antagonist; CS-3150; Japanese
MeSH Terms: conditions — Essential Hypertension | interventions — esaxerenone; Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- CS-3150 1.25 mg (Experimental): One CS-3150 1.25 mg tablet and one placebo tablet to match CS-3150 tablet administered orally, once daily after breakfast.
  Interventions: Drug: CS-3150; Drug: placebo
- CS-3150 2.5 mg (Experimental): Two CS-3150 1.25 mg tablets administered orally, once daily after breakfast.
  Interventions: Drug: CS-3150
- CS-3150 5 mg (Experimental): Two CS-3150 2.5 mg tablets administered orally, once daily after breakfast.
  Interventions: Drug: CS-3150
- Placebo (Placebo Comparator): Two placebo tablets to match CS-3150 tablet, administered orally, once daily after breakfast.
  Interventions: Drug: placebo
- Eplerenone, 50-100 mg (Open Label) (Active Comparator): One or two 50mg eplerenone tablet(s) administered orally, once daily after breakfast.
  Interventions: Drug: eplerenone

INTERVENTIONS:
Drug: CS-3150
  Arms: CS-3150 1.25 mg; CS-3150 2.5 mg; CS-3150 5 mg
Drug: placebo
  Arms: CS-3150 1.25 mg; Placebo
Drug: eplerenone
  Arms: Eplerenone, 50-100 mg (Open Label)

SUMMARY:
This study is a randomized, placebo-controlled, double-blind, multi-center study to evaluate efficacy and safety of different doses of CS-3150 compared to placebo in Japanese hypertensive subjects. Primary endpoint is change from baseline in sitting systolic and diastolic blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 20 years or older at informed consent
* Subjects with essential hypertension (Sitting SBP ≥ 140 mmHg and < 180 mmHg, Sitting DBP ≥ 90 mmHg and < 110 mmHg,and 24h-hr blood pressure more than 130 mmHg in SBP and 80 mmHg in DBP)

Exclusion Criteria:

* Secondary hypertension or malignant hypertension
* Diabetes mellitus with albuminuria
* Serum potassium level < 3.5 or ≥ 5.1 mEq/L
* Reversed day-night life cycle including overnight workers
* eGFR < 60 mL/min/1.73 m^2

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sitting systolic and diastolic blood pressure | baseline to end week 12

SECONDARY OUTCOMES:
Change from baseline in 24-hr blood pressure (ABPM) | Baseline to end week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/